CLINICAL TRIAL: NCT02792582
Title: A Phase II Trial of Intensity-Modulated Proton Therapy for Incompletely Resected Craniopharyngioma and Observation for Craniopharyngioma After Radical Resection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT3CR; NCI-2016-00813 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Craniopharyngioma
Keywords: Brain tumor; Pediatrics; Radiation therapy; Proton therapy; Surgery
MeSH Terms: conditions — Craniopharyngioma; Brain Neoplasms | interventions — Proton Therapy; Radiotherapy; Surgical Procedures, Operative; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Tumor-Surgery (Active Comparator): Participants who are eligible to undergo surgery to remove the tumor will proceed to surgery. If all tumor is removed, they will be followed over 5 years for outcome comparison to the other participant groups.
  If the entire tumor is not removed by surgery, participants will receive 6 weeks of proton therapy. They will then be followed for 5 years to collect outcome data for comparison to the other participant groups.
  Interventions: Radiation: Proton Therapy; Procedure: Surgery
- Tumor-No Surgery (Active Comparator): Participants whose tumor cannot be resected through surgery will receive 6 weeks of proton therapy. They will then be followed over 5 years for outcome comparison to the other participant groups.
  Interventions: Radiation: Proton Therapy

INTERVENTIONS:
Radiation: Proton Therapy — The protocol-specific radiation dose will be prescribed to a target defined by the use of computerized tomography (CT) and magnetic resonance imaging (MRI). The target will encompass the residual tumor and/or tumor bed and will include a margin mean to treat subclinical microscopic disease. There is no time limit for the interval from surgery or study enrollment to when proton therapy commences. The time course of administration of proton therapy will be 1 treatment/day, 5 days/week, for a period 6 weeks.
  Other Names: Radiation therapy
Procedure: Surgery — When possible, tumors will be removed surgically prior to proton therapy. If no tumor remains following surgery, no proton therapy will be given, and participants will be followed for 5 years to collect outcome data for comparison between groups.
  Other Names: Tumor resection
  Arms: Tumor-Surgery

SUMMARY:
Craniopharyngioma is a rare brain tumor that affects both children and adults. It arises in a region of the brain near the pituitary gland, visual pathways, and central blood vessels. Patients often present with headache, loss of vision or delayed growth. In some instances they may present with imbalance of water and salts in the body.

The treatment for craniopharyngioma may be radical surgery or a combination of surgery and radiation therapy. In some instances surgery is not required. If the tumor cannot be completely removed, radiation therapy may be required. In this study we will use the most advanced form of proton therapy which is called intensity-modulated proton therapy. This is a newer form of radiation therapy which has a number of advantages over older forms of proton therapy and conventional radiation therapy using x-rays.

The main goal of this study is to learn if proton therapy will effectively treat patients with craniopharyngioma brain tumors and reduce side effects compared to more traditional forms of radiation therapy.

DETAILED DESCRIPTION:
This study will include participants who are diagnosed or presumed to have craniopharyngioma based on neuroimaging, intra-operative assessment, or the evaluation of cyst fluid or tissue after limited or radical surgery. When possible, participants will be enrolled on protocol prior to surgery.

PRIMARY OBJECTIVE:

* To estimate the distributions of progression-free and overall survival for children and young adults with craniopharyngioma treated with intensity-modulated proton therapy while monitoring for excessive central nervous system necrosis, clinically significant vasculopathy, and permanent neurological conditions or deficits.

SECONDARY OBJECTIVES:

* To estimate the cumulative incidence of cystic intervention and the event-free survival distribution for children and young adults with craniopharyngioma treated with intensity-modulated proton therapy; and to compare the distributions of progression-free, event-free and overall survival with the distributions for the St. Jude Children's Research Hospital (SJCRH) cohort of patients treated with photon therapy on which the design of this trial is based.
* To estimate the cumulative incidence of cystic intervention and the distributions of progression-free survival, overall survival and the event-free survival for children and young adults with craniopharyngioma treated only with primary surgical resection and to compare these distributions with the distributions observed for patients treated with proton therapy.

OTHER PRE-SPECIFIED OBJECTIVES:

* To explore potential associations of clinical and treatment factors with the incidence and severity of neurological, endocrine and cognitive deficits in children and young adults with craniopharyngioma treated with radical surgery or proton therapy. Descriptively compare findings for patients treated with proton therapy with the reported findings for the updated SJCRH cohort treated with photon therapy.
* Using specific measures of sleep quality, excessive daytime sleepiness, daytime activity, circadian rhythm, fatigue, symptom distresses, and quality of life, explore associations of sleep, fatigue and quality of life with other measures of central nervous system (CNS) effects, clinical and treatment factors in children and young adults with craniopharyngioma treated with radical surgery or proton therapy.
* To evaluate and explore differences in physical performance and movement in children and young adults with craniopharyngioma treated with radical surgery or proton therapy, using specific measures of overall physical performance, flexibility, balance, coordination, muscle strength and power, and cardiopulmonary fitness.
* Estimate and compare the response of residual tumor and the incidence and severity of structural, functional and vascular effects of normal brain in children and young adults with craniopharyngioma after treatment with radical surgery or proton therapy using specific methods of diffusion, contrast-enhancement, vascular and functional neuroimaging, and explore the association between these and other measures of CNS effects and clinical and treatment factors.
* Investigate the feasibility of using positron emission tomography (PET) as an in vivo dose and distal edge verification system for craniopharyngioma patients treated with proton therapy.
* Measure growth factor and cytokine responses in children and young adults with craniopharyngioma after treatment with radical surgery or proton therapy, and explore associations between these and other measures of CNS effects and clinical and treatment factors. Descriptively compare findings for patients treated with proton therapy with the reported findings for the updated SJCRH cohort treated with photon therapy.

ELIGIBILITY:
Inclusion Criteria:

* Craniopharyngioma diagnosed by histology, cytology or neuroimaging or intra-operative assessment
* Patients ages 0-21 years at the time of diagnosis

Exclusion Criteria:

* Prior history of fractionated radiation therapy
* Prior treatment with intracystic P-32 or intracystic bleomycin
* Pregnant females are excluded. Radiation has teratogenic or abortifacient effects

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 years after initiation of proton therapy
  PFS is defined as the interval of time from the initiation of radiation therapy (RT) until the earliest of the events: death from any cause; and disease progression.
Overall survival (OS) | 3 years after initiation of proton therapy
  OS is defined as the interval of time from the initiation of RT until the death from any cause.

SECONDARY OUTCOMES:
Compare incidence of first cystic intervention with participants treated with conventional radiation therapy at St. Jude Children's Research Hospital | 3 years after initiation of proton therapy
  The cumulative incidence estimates of first cystic intervention for cystic fluctuations after proton therapy. Competing events are death, disease progression and development of a new or secondary tumor.
Compare event-free survival (EFS) with participants treated with conventional radiation therapy at St. Jude Children's Research Hospital | 3 years after initiation of proton therapy
  Kaplan-Meier estimates will be provided of EFS, which is measured from initiation of proton therapy until the earliest of PFS failure or secondary malignancy or new tumor, or surgical intervention for cystic fluctuation. Patients who have not experienced an event will be censored at their last date of contact.
Compare survival distributions with participants treated with conventional radiation therapy at St. Jude Children's Research Hospital | 3 years after initiation of proton therapy
  Final analyses will also compare survival distributions using the log-rank test for patients treated with limited surgery and proton therapy on this protocol with the updated SJCRH cohort of patients treated with limited surgery and photon irradiation. The definition of survival will be defined in same way for both cohorts. This secondary analysis will be stratified by whether or not patients have a cerebrospinal fluid (CSF) shunt in place prior to irradiation and race (black versus white).
Compare survival distributions between groups | 3 years after initiation of proton therapy
  To estimate the survival distributions for children and young adults with craniopharyngioma treated only with primary surgical resection and to compare these distributions with the distributions observed for patients treated with limited surgery and proton therapy. A stratified log-rank test will be used to compare the distributions for children and young adults with craniopharyngioma treated only with primary surgical resection and the distributions observed for patients treated with limited surgery and proton therapy.

OTHER OUTCOMES:
Change in vision status compared between groups | From baseline to 5 years following start of proton therapy
  Vision status will be classified into three groups (None, Impaired, Severe). Information recorded in the clinical neurology form will also be used, as will the ophthalmology data sheet and NCI CTCAE v4.0 when relevant. The distribution of outcomes is ordinal categorical and percentages will be estimated. Mixed-effects Proportional Odds Regression will be used to estimate the change of vision over time, and compare severity of vision in the two treatment groups adjusted by confound factors.
Change in hearing status compared between groups | From baseline to 5 years following start of proton therapy
  Hearing will be categorized as normal if all thresholds are within 0-20 decibels hearing level (dB HL) and otherwise abnormal. Generalized Estimating Equations (GEE) with logistic link will be used to explore the trend over time and investigate impacts of specific clinical and treatment factors on hearing loss. In the presence of missing data, Weighted GEE will be employed to address missingness. In addition, the cumulative incidence of hearing loss will be estimated with death as a competing risk.
Compare number of neurological deficits to participants treated using conventional radiation therapy at St. Jude Children's Research Hospital | From baseline to 5 years following start of proton therapy
  The incidence and severity of neurological deficits in children and young adults with craniopharyngioma treated with radical surgery or limited surgery and proton therapy. Descriptively compare findings for patients treated with proton therapy with the reported findings for the updated SJCRH cohort treated using photons.
Compare number of endocrine deficits to participants treated using conventional radiation therapy at St. Jude Children's Research Hospital | From baseline to 5 years following start of proton therapy
  The incidence and severity of endocrine deficits in children and young adults with craniopharyngioma treated with radical surgery or limited surgery and proton therapy. Descriptively compare findings for patients treated with proton therapy with the reported findings for the updated SJCRH cohort treated using photons.
Compare number of cognitive deficits to participants treated using conventional radiation therapy at St. Jude Children's Research Hospital | From baseline to 5 years following start of proton therapy
  The incidence and severity of cognitive deficits in children and young adults with craniopharyngioma treated with radical surgery or limited surgery and proton therapy. Descriptively compare findings for patients treated with proton therapy with the reported findings for the updated SJCRH cohort treated using photons.
Compare quality of life between groups | From baseline to 5 years following start of proton therapy
  Analysis will be stratified by treatment arms (radical surgery vs. limited surgery and proton therapy), descriptive statistics of the longitudinal assessments of quality of life will be described. Specifically, on a yearly basis starting from the pre-treatment time point to year 5 post treatment initiation, quality of life in patients ≥ 2 years of age as measured by the Peds QoL v4 and the Peds QoL brain tumor module will be reported. On a more frequent basis (every 3 months in the first year after treatment initiation and every 6 months afterwards), sleep complaints in patients ≥ 8 years of age as measured Epworth Sleepiness Scale will be reported and fatigue in patients ≥ 2 years of age as measured by The Peds QL Multidimensional Fatigue scale will be reported. Sleep disorders at diagnosis and 3 years after the initiation of treatment will be measured by overnight polysomnography.
Compare physical performance and movement between groups | From baseline to 5 years following start of proton therapy
  Physical performance measures will be obtained at baseline, 6, 12, 24, 36, 48 and 60 months. For the surgery only group, baseline is measured immediately after surgery. For the limited surgery and proton therapy group, the baseline is measured immediately before proton therapy. The baselines in the two groups are measured approximately at the same time so the comparisons between the two groups are reasonable. Descriptive statistics of the outcomes for each group will be provided.
Incidence of vasculopathy between groups | From baseline to 5 years following start of proton therapy
  Cumulative incidence of vasculopathy with at least major symptoms (i.e., Vasculopathy grade > 2) will be estimated for the first occurrence of vasculopathy, where death, disease progression, and development of a new or secondary tumor will be considered as completing events. Vasculopathy will be graded 3-5 according to NCI CTCAE v4.0.
Compare incidence of central nervous effects between groups | From baseline to 5 years following start of proton therapy
  Quantitative measures of structural and functional changes in the brain over time will be described using mixed effects models. Associations of functional and structural changes in the brain with cognitive variables will be investigated using mixed effects models which will include demographic, imaging and clinical factors, such as age at diagnoses, gender, race and socioeconomic status, fractional anisotropy (FA), apparent diffusion coefficient (ADC), hydrocephalus and presence of CSF shunt, and pre-proton therapy growth hormone deficiency.
Percentage of participants who were successfully evaluated with an in vivo dose and distal edge verification system | From baseline to 5 years following start of proton therapy
  The percentage of patients with PET scans where loss of signal intensity or resolution was observed will be estimated with 95% exact confidence intervals.
Change in growth factor response | From baseline to 5 years following start of proton therapy
  The planned analyses based on this data will mainly utilize longitudinal models.
Change in cytokine response | From baseline to 5 years following start of proton therapy
  The planned analyses based on this data will mainly utilize longitudinal models.
Number and type of germline variations associated with craniopharyngioma | 5 years following start of proton therapy
  Descriptive statistics will be provided for known candidate genes and gene mutations. Analysis will be performed using current processes available at the time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Merchant, DO, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Wilson LJ, Pirlepesov F, Moskvin V, Li Z, Guo Y, Li Y, Merchant TE, Faught AM. Proton therapy delivery method affects dose-averaged linear energy transfer in patients. Phys Med Biol. 2021 Apr 1;66(7). doi: 10.1088/1361-6560/abe835. PMID 33607632
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols